CLINICAL TRIAL: NCT01861431
Title: Evaluating a Microfinance Intervention for High Risk Women in Mongolia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Witte, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAF4402; R34MH093227 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infection
Keywords: HIV, prevention, microfinance, sex work, Mongolia
MeSH Terms: conditions — HIV Infections; Sex Work

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIVSRR (Active Comparator): 4 sessions of HIV sexual risk reduction
  Interventions: Behavioral: HIV Sexual Risk reduction
- HIVSRR + Microfinance (Experimental): 4 sessions of sexual risk reduction plus 12 sessions of financial literacy, 12 sessions of business development training, 10 sessions of business mentorship; matched savings throughout course of intervention
  Interventions: Behavioral: HIV Sexual Risk reduction plus Microfinance

INTERVENTIONS:
Behavioral: HIV Sexual Risk reduction — 4 sessions of HIV sexual risk reduction
  Arms: HIVSRR
Behavioral: HIV Sexual Risk reduction plus Microfinance — 4 sessions of sexual risk reduction plus 12 sessions of financial literacy, 12 sessions of business development training, 10 sessions of business mentorship; matched savings throughout course of intervention
  Arms: HIVSRR + Microfinance

SUMMARY:
The proposed study aims to test the feasibility and preliminary efficacy of a combined 4-session HIV sexual risk reduction (HIVSRR) and microfinance intervention (including 34 training session and matched savings) to reduce unprotected sex and to increase proportion of income from sex work among women engaged in high risk sexual activity in Ulaanbaatar, Mongolia. Feasibility and preliminary efficacy will be tested using a randomized clinical trial (RCT) with 134 women sex workers meeting eligibility criteria. Following eligibility screening, eligible women will complete informed consent, a baseline assessment, and be randomized to one of 2 study conditions: 1) the combination HIV sexual risk reduction plus microfinance (HIVSRR+MF); or 2) a 4-session HIVSRR alone control condition.

The study design will permit us to:

1. Examine and enhance the feasibility (i.e. recruitment, engagement, attendance, retention data collection) of a combination HIV sexual risk reduction and MF intervention with high risk women in Ulaanbaatar, Mongolia;
2. Examine the preliminary outcomes of the interventions on decreasing unprotected acts of vaginal and anal intercourse; increasing the proportion of protected vaginal and/or anal acts using barrier protection and decreasing number of sexual partners with repeated measures at baseline, immediately post-intervention, and 3 and 6 month follow-up assessments.
3. Use the results of the pilot study to inform the design of a future R01 application.

ELIGIBILITY:
Inclusion Criteria:

* She is at least 18 years of age;
* She reports having engaged in vaginal or anal sexual intercourse in the past 90 days in exchange for money, alcohol or other goods;
* She reports having engaged in unprotected vaginal or anal sexual intercourse in the past 90 days with a paying sexual partner; and
* She reports being interested in learning about and developing her own small business.

Exclusion Criteria:

* assessed to have a severe cognitive or psychiatric impairment that would interfere with the ability to provide informed consent or complete study instruments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
unprotected acts of vaginal and anal intercourse; | 6 months
  The primary outcomes include: decreasing unprotected acts of vaginal and anal intercourse; increasing the proportion of protected vaginal and/or anal acts using barrier protection and decreasing number of sexual partners with repeated measures at baseline, immediately post-intervention, and 3 and 6 month follow-up assessments.

SECONDARY OUTCOMES:
proportion of protected vaginal and/or anal acts using barrier protection; | 6 months
number of sexual partners | 6 months
Proportion of income from sex work | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Witte, PhD, Principal Investigator — Columbia University
Locations (1):
- Aira Toivgoo, co-PI, Ulaanbaatar, Mongolia

REFERENCES:
- [Derived] Tsai LC, Carlson CE, Aira T, Norcini Pala A, Riedel M, Witte SS. The impact of a microsavings intervention on reducing violence against women engaged in sex work: a randomized controlled study. BMC Int Health Hum Rights. 2016 Oct 28;16(1):27. doi: 10.1186/s12914-016-0101-3. PMID 27793147